CLINICAL TRIAL: NCT01900197
Title: A Non-intervention Trial of the Time to Relapse of Iron Deficiency Anemia After Standard Treatment With a New Intravenous Iron (Monofer®)
Brief Title: Time to Relapse of Iron Deficiency Anemia After Standard Treatment With a New Intravenous Iron (Monofer®)
Status: Completed | Type: Observational
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: BioStata (Industry)
Responsible Party: Sponsor
Other Study IDs: Monofer®-NIS-14
Record Dates: First submitted 2013-07-11; First posted 2013-07-16 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — iron isomaltoside 1000

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Iron deficiency anemia: Patients with iron deficiency anemia treated on the doctor's discretion with 10% Iron Isomaltoside 1000 (Monofer®) as standard treatment according to current practice
  Interventions: Drug: 10% Iron Isomaltoside 1000

INTERVENTIONS:
Drug: 10% Iron Isomaltoside 1000 — Administered according to local routines and product labeling in doses at the doctors discretion
  Other Names: Monofer®

SUMMARY:
The purpose of this study is to monitor and quality assure the efficacy and safety of Monofer® in a broad patient population when Monofer® is used according to the Monofer® label (SPC) in current practice and where standard routines are being followed.

DETAILED DESCRIPTION:
The total duration of the study is approximately 21 months, which includes a 6 months enrolment period. The number of patient visits depends on the number of Monofer® treatment courses needed during the study period. Each patient can receive one or more treatment courses during 12 months after informed consent. The last blood test will be taken after the last Monofer® treatment course which might occur 13-15 months after Informed consent. Patients will only attend hospital visits planned as part of their standard treatment and they will receive treatment as a part of standard care and according to the doctor's discretion. Study termination will occur once the 12 months observational period has been completed for all patients and the last blood test has been collected from the last Monofer® treated patient in the study. Each treatment course can consist of one or more Monofer® administrations. For each administration of Monofer® either intravenous infusion or injection can be used. Pre- and post-treatment blood tests according to standard treatment are a part of the Monofer® treatment course.

DATA COLLECTION:

* Clinical data management will be performed in accordance with applicable standards and data cleaning procedures.
* The collected data will systematically be entered into an eCRF (MyEDC, Biostata). The source of information is the relevant laboratory results obtained from the patient record.
* The data will be evaluated by the Pharmacosmos A/S Medical Affairs team.

Laboratory assessments, i.e. anemia work-up/treatment evaluation, shall be a part of local standard practice. The protocol does not accept any additional samples outside current local standard practice to be taken.

ELIGIBILITY:
Inclusion Criteria:

Patients with iron deficiency anemia treated on the doctor's discretion with Monofer® as standard treatment according to current practice

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with iron deficiency anemia treated on the doctor's dicretion with Monofer® as standard treatment according to current practice
Sampling Method: Probability Sample
Enrollment: 391 (Actual)
Dates: Start 2013-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Time to relapse of iron deficiency anemia | From screening until 12 months

SECONDARY OUTCOMES:
Number of ADRs | From screening until 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg, Denmark

REFERENCES:
- [Derived] Frigstad SO, Haaber A, Bajor A, Fallingborg J, Hammarlund P, Bonderup OK, Blom H, Rannem T, Hellstrom PM. The NIMO Scandinavian Study: A Prospective Observational Study of Iron Isomaltoside Treatment in Patients with Iron Deficiency. Gastroenterol Res Pract. 2017;2017:4585164. doi: 10.1155/2017/4585164. Epub 2017 Oct 22. PMID 29213281